CLINICAL TRIAL: NCT05205018
Title: Remote Motivational Interviewing to Improve Self-care in Heart Failure Patients
Acronym: ReMotivateHF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Ercole Vellone, Associate Professor, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 263/21
Record Dates: First submitted 2022-01-09; First posted 2022-01-24 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Heart Failure
Keywords: heart failure; motivational interviewing; self-care; self-management; behavior change; Video calls
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing Arm (Experimental): This Arm will receive a remote intervention (via videacalls) based on motivational interviewing to improve self-care. The intervention will be delivered seven time over 12 months.
  Interventions: Behavioral: Motivational interviewing performed remotely through videocalls
- Standard care Arm (No Intervention): This Arm will receive the standard of care.

INTERVENTIONS:
Behavioral: Motivational interviewing performed remotely through videocalls — Remote motivational interviewing will be performed seven time over 12 months, through videocalls. The first four interventions will be performed within two months and the following three will be performed at five, eight and eleven months from enrollment.
  Arms: Motivational Interviewing Arm

SUMMARY:
The purpose of this study is to evaluate if motivational interviewing, performed remotely through videocalls, is effective to improve self-care in patients with heart failure

DETAILED DESCRIPTION:
After signing the informed consent form, patients with heart failure will be assigned to the intervention or control group (1:1). The intervention group will receive a total of seven motivational interviewing sessions over 12 months. The control group will receive the standard care.

ELIGIBILITY:
Inclusion Criteria:

1. a diagnosis of HF according to international guidelines;
2. Class II, III or IV in the New York Heart Association (NYHA) functional;
3. poor self-care, defined as at least two items of the Self-Care Heart Failure Index 7.2 (SCHFI 7.2) with a score of 0, 1 or 2;
4. age ≥ 18 years;
5. having an internet access to allow the videocalls;
6. willingness to sign the informed consent form. -

Exclusion Criteria:

1. severe cognitive dysfunction, with a score 0 - 4 on the Six-item screener;
2. acute coronary events event in the prior three months;
3. living in nursing homes a residential settings where self-care cannot be performed;
4. if the patient's informal caregiver is not willing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Self-care maintenance | 3 months from enrollment
  Self-care maintenance will be measured with the Self-Care Maintenance Scale of the Self-Care of Heart Failure Index v.7.2

SECONDARY OUTCOMES:
Self-care maintenance | 6, 9 and 12 months from enrollment
  Self-care maintenance will be measured with the Self-Care Maintenance Scale of the Self-Care of Heart Failure Index v.7.2
Self-care monitoring | 3, 6, 9 and 12 months from enrollment
  Self-care monitoring will be measured with the Self-Care Monitoring Scale of the Self-Care of Heart Failure Index v.7.2
Self-care management | 3, 6, 9 and 12 months from enrollment
  Self-care monitoring will be measured with the Self-Care Management Scale of the Self-Care of Heart Failure Index v.7.2
Self-Care Self-Efficacy levels | 3, 6, 9 and 12 months from enrollment
  Self-Care Self-Efficacy will be measured with the Self-Care Self-Efficacy Scale; this scale gives a score from 0 to 100 with higher score meaning higher self-care self-efficacy
Burden of heart failure physical symptoms | 3, 6, 9 and 12 months from enrollment
  The burden of heart failure physical symptom will be measured with the Heart Failure Somatic Perception Scale
Disease specific quality of life | 3, 6, 9 and 12 months from enrollment
  The disease-specific quality of life will be measured with the Kansas City Cardiomyopathy Questionnaire
Caregiver contribution to heart failure self-care | 3, 6, 9 and 12 months from enrollment
  Will be evaluated with the Caregiver Contribution to Self-Care of Heart Failure Index 2
Caregiver preparedness | 3, 6, 9 and 12 months from enrollment
  Will be evaluated with the Caregiver Preparedness Scale
Caregiver burden | 3, 6, 9 and 12 months from enrollment
  Will be evaluated with the Caregiver Burden Inventory
Health care service uses | 3, 6, 9 and 12 months from enrollment
  They will be evaluated with a questionnaire developed by the research team. Specifically wi will evaluate patient mortality, hospitalizations and used of emergency services.
Patient and caregiver generic quality of life | 3, 6, 9 and 12 months from enrollment
  Generic quality of live in patients and in caregivers will be evaluated with the SF-12 Survey
Patient and caregiver anxiety and depression | 3, 6, 9 and 12 months from enrollment
  They will ve evaluated with the Hospital Anxiety and Depression Scale
Naturalistic decision making of patients and caregivers | 3, 6, 9 and 12 months from enrollment
  They will be evaluated with the Naturalistic Decision Making Scale (patient and caregiver version)

CONTACTS AND LOCATIONS:
Overall Officials: Ercole Vellone, PhD, Principal Investigator — University of Rome Tor Vergata
Locations (1):
- Hospital of Alessandria, Alessandria, Italy

IPD SHARING:
Plan to Share IPD: No